CLINICAL TRIAL: NCT00003104
Title: A Phase II Study Using High Dose Three Dimensional Conformal Radiation Therapy in Intermediate Prognostic Risk Patients With Adenocarcinoma of the Prostate
Brief Title: Computer Planned Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 97-064; CDR0000065838 (Registry Identifier: PDQ (Physician Data Query)); NCI-H97-0006
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Computer systems that allow doctors to create a 3-dimensional picture of the tumor in order to plan treatment may result in more effective radiation therapy.

PURPOSE: This phase II trial is studying how well radiation therapy that has been planned with a computer works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish the efficacy of high-dose three-dimensional conformal radiotherapy in patients with intermediate prognostic risk adenocarcinoma of the prostate.
* Determine the PSA relapse-free survival rate of this patient population.

OUTLINE: Patients receive high-dose three-dimensional conformal radiotherapy 4-5 days per week for at least 9 weeks.

Patients are evaluated at least weekly during radiotherapy and at 2 and 4 months after treatment completion. Thereafter, patients are followed every 6 months for a total of 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven intermediate prognostic risk (T1-T2) adenocarcinoma of the prostate

  * Previously untreated (except for hormonal therapy)
  * PSA levels greater than 10 ng/mL and Gleason scores no greater than 6 OR
  * PSA levels no greater than 10 ng/mL and Gleason scores at least 7
  * Patients requiring volume reduction of prostate prior to radiotherapy continue to be treated at least 3 months on neoadjuvant hormonal therapy prior to radiation
* No evidence of distant metastases
* No regional lymph node involvement

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No major medical illness
* No psychosis
* No metallic pelvic prosthesis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Prior neoadjuvant antiandrogen therapy allowed

Radiotherapy:

* No prior radiotherapy
* No prior pelvic irradiation

Surgery:

* No prior radical surgery for carcinoma of the prostate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1997-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Zelefsky, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States